CLINICAL TRIAL: NCT00751023
Title: Effects of Modafinil in Methamphetamine Dependence
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HR#18440
Record Dates: First submitted 2008-09-10; First posted 2008-09-11 (Estimated); Results first posted 2019-06-13 (Actual); Last update posted 2019-06-13 (Actual); Status verified 2019-05

CONDITIONS: Methamphetamine Dependence
Keywords: Methamphetamine; Modafinil; Addiction; Craving; Cognitive
MeSH Terms: conditions — Behavior, Addictive | interventions — Modafinil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Modafinil 400 mg daily
  Interventions: Drug: Modafinil
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Modafinil — 400 mg daily for four weeks
  Other Names: Provigil
  Arms: 1
Drug: Placebo — Placebo 2 tablets daily for 4 weeks
  Arms: 2

SUMMARY:
Methamphetamine dependence is a serious public health problem with no pharmacologic treatments currently available. Relapse rates are high in this population. Exposure to cues previously associated with methamphetamine use may induce profound craving in abstinent individuals. Chronic methamphetamine abuse is associated with selective cognitive deficits that may undermine successful participation in psychosocial treatments. Medications which improve cognitive deficits in methamphetamine-dependent individuals may improve abstinence rates, especially in the critical early period of recovery. Modafinil is an atypical stimulant medication with evidence to support its use in treating cocaine dependence and attention deficit/hyperactivity disorder. The proposed studies are designed to evaluate modafinil as a potential treatment for methamphetamine dependence and its cognitive sequelae.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be able to provide informed consent and function at an intellectual level sufficient to allow accurate completion of all assessment instruments.
2. Subjects must meet DSM-IV criteria for methamphetamine dependence within the past six months. Subjects may meet criteria for abuse, but not dependence on any other substance with the exception of nicotine. Because of the high comorbidity of methamphetamine and nicotine dependence, excluding nicotine dependence would seriously compromise the feasibility of recruitment. Nicotine use immediately prior to the cue reactivity testing session will be controlled.
3. Subjects must consent to remain abstinent from all drugs of abuse (except nicotine) for 24 hours prior to the cue reactivity testing sessions.
4. Subjects must consent to random assignment to the modafinil vs. placebo conditions.

Exclusion Criteria:

1. Women who are pregnant, nursing or of childbearing potential and not practicing an effective means of birth control.
2. Subjects with evidence of or a history of significant hematological, endocrine, cardiovascular, pulmonary, renal, gastrointestinal, or neurological disease as these conditions may affect heart rate or skin conductance measurement.
3. Subjects with a history of or current psychotic disorder or bipolar affective disorder as these may impact cue reactivity.
4. Subjects who are unwilling or unable to maintain abstinence from alcohol and other drugs of abuse (except nicotine) for 24 hours prior the cue procedures.
5. Subjects meeting DSM-IV criteria for substance dependence (other than nicotine or methamphetamine as appropriate) within the past 60 days.
6. Subjects currently taking B-blockers, anti-arrhythmic agents, psychostimulants or any other agents known to interfere with heart rate and skin conductance monitoring.
7. Known or suspected hypersensitivity to modafinil.
8. Individuals taking medications that could adversely interact with study medications.
9. Subjects with a history of epilepsy or seizure disorder.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-02; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bryan K Tolliver, MD, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Behavioral Health Services of Pickens County, Pickens, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The Enrollment number in the Protocol Section has been corrected (n=40) to appropriately match the number of participants listed in the Results Participant Flow section. The previous Protocol section incorrectly included a cohort (n=31) of healthy control subjects who underwent cognitive testing but did not participate in the modafinil trial.
Groups:
- Modafinil: Modafinil 400 mg daily
  Modafinil: 400 mg daily for four weeks
- Placebo: Placebo
  Placebo: Placebo 2 tablets daily for 4 weeks
Period: Overall Study
Arm/Group | Modafinil | Placebo
Started | 20 | 20
Completed | 9 | 13
Not Completed | 11 | 7
Not completed — Lost to Follow-up | 11 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Modafinil | Placebo | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.3 (8.2) | 32.1 (7.4) | 31.2 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 27
  Male | 6 | 7 | 13

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Methamphetamine-positive Urine Drug Screens
Description: Percentage of participants with at least one biweekly urine drug screen positive for methamphetamine (4 weeks active treatment phase + medication-free safety visit at week 5)
Time Frame: 5 weeks
Measure: Number; unit: Percentage of participants
Arm/Group | Modafinil | Placebo
Number analyzed (Participants) | 20 | 20
Percentage of participants | 85 | 65

2. Secondary Outcome: Percent Change in California Verbal Learning Test From Baseline to Study Endpoint
Description: Mean percent change in T scores (average total score of 6 trials) from baseline to study endpoint (Week 5) in study completers. Larger (more positive) percent change values indicate better outcomes.
Time Frame: Study baseline to study endpoint (Week 5)
Measure: Mean (Standard Deviation); unit: Percent change, baseline-study endpoint
Arm/Group | Modafinil | Placebo
Number analyzed (Participants) | 9 | 13
Percent change, baseline-study endpoint | 20.6 (13.4) | 14.8 (4.9)

3. Secondary Outcome: Percent Change in Symbol Digit Modalities Test From Baseline to Study Endpoint
Description: Mean percent change in T scores from baseline to study endpoint (Week 5) in study completers. Larger (more positive) percent change values indicate better outcomes.
Time Frame: 5 Weeks
Measure: Mean (Standard Deviation); unit: Percent change, baseline-study endpoint
Arm/Group | Modafinil | Placebo
Number analyzed (Participants) | 9 | 13
Percent change, baseline-study endpoint | 6.4 (15.2) | 10.0 (23.6)

4. Secondary Outcome: Percent Change in Paced Auditory Serial Addition Test Scores From Baseline to Study Endpoint
Description: Mean percent change of T scores from baseline to study endpoint (Week 5) in study completers. Min T score = 0, max T score = 100. Higher scores, greater (more positive) percent change indicate better outcomes.
Time Frame: 5 weeks
Measure: Mean (Standard Deviation); unit: Percent change, baseline-study endpoint
Arm/Group | Modafinil | Placebo
Number analyzed (Participants) | 9 | 13
Percent change, baseline-study endpoint | 11.3 (23.5) | 28.5 (61.0)

5. Secondary Outcome: Score on the Wisconsin Card Sort Test
Description: Scores (T scores) on the Wisconsin Card Sort Test (total errors) at study endpoint (Week 5) in study completers, adjusted for age and education; min=0, max=100, higher numbers indicate better outcomes.
Time Frame: 5 weeks
Population: Note: Total number of study completers = 22 (9 in Modafinil group and 13 in Placebo group). The Wisconsin Card Sort Test was able to be completed in only 19 of 22 study completers (8 participants assigned to Modafinil and 11 participants assigned to Placebo).
Measure: Mean (Standard Deviation); unit: T scores at study endpoint
Arm/Group | Modafinil | Placebo
Number analyzed (Participants) | 8 | 11
T scores at study endpoint | 44.6 (14.0) | 41.9 (14.5)

6. Secondary Outcome: Percent Change in the Grooved Pegboard Test Score From Baseline to Study Endpoint
Description: Percent change of T scores from baseline to study endpoint (Week 5) in study completers; T score min=0, max=100; higher scores (more positive change) indicate better outcome.
Time Frame: 5 weeks
Measure: Mean (Standard Deviation); unit: Percent change, baseline-study endpoint
Arm/Group | Modafinil | Placebo
Number analyzed (Participants) | 9 | 13
Percent change, baseline-study endpoint | 10.8 (40.7) | 65.0 (149.9)

7. Secondary Outcome: Percent Change in Shipley Institute of Living Scale Scores From Baseline to Study Endpoint
Description: Percent change in scores (T scores) on the Shipley Abstract subscale from baseline to study endpoint (Week 5) in study completers; T scores min=0, max=100; larger positive values indicate better outcome.
Time Frame: 5 weeks
Measure: Mean (Standard Deviation); unit: T scores, percent change
Arm/Group | Modafinil | Placebo
Number analyzed (Participants) | 9 | 13
T scores, percent change | 4.1 (7.1) | 4.6 (16.3)

8. Secondary Outcome: Percentage Change in Beck Depression Inventory Scores
Description: Percent change in BDI score from baseline to study endpoint in study completers; range =-100% to 100%, larger (more negative) change indicates better outcome.
Time Frame: 5 weeks
Population: Note: Total number of study completers = 22 (9 in Modafinil group and 13 in Placebo group). Beck Depression Inventory Scores at study endpoint were obtained in only 20 of 22 study completers (9 participants assigned to Modafinil and 11 participants assigned to Placebo).
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Modafinil | Placebo
Number analyzed (Participants) | 9 | 11
Percent change | -58.4 (52.7) | -43.5 (35.4)

ADVERSE EVENTS:
Time Frame: Five weeks: Four weeks of active study medication, safety visit one week after medication washout
Description: Adverse events were systematically collected using a standardized questionnaire at each semi-weekly visit (9 visits total over 5 weeks)
Groups:
- Placebo: Placebo: 2 tablets daily for four weeks
Arm/Group | Modafinil | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 16/20 | 14/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Modafinil (N=20) | Placebo (N=20)
Anxiety (Psychiatric disorders) | 5 (5) | 2 (2)
Nausea (Gastrointestinal disorders) | 4 (4) | 2 (2)
Insomnia (General disorders) | 2 (2) | 3 (3)
Headache (General disorders) | 4 (4) | 1 (1)
Common cold symptoms (General disorders) | 2 (2) | 3 (3)
Hypersomnia (General disorders) | 2 (2) | 3 (3)
Abdominal cramps (Gastrointestinal disorders) | 0 (0) | 4 (4)
Decreased appetite (General disorders) | 3 (3) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Dry mouth / thirst (General disorders) | 2 (3) | 1 (1)
Ear / sinus infection (Infections and infestations) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Elevated blood pressure (General disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
Limited sample size (n=40, n=20 in each group), relatively low retention (55% overall; 45% in modafinil group, 65% in placebo group)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No